CLINICAL TRIAL: NCT05437744
Title: Assessment of Soft Tissue Healing Over Immediately Placed Implant Sealed With Platelets Rich Fibrin (Prf) Versus Cyanoacrylate Glue (a Randomized Controlled Clinical Trial)
Brief Title: Immediately Placed Implant Sealed With Platelets Rich Fibrin Versus Cyanoacrylate Glue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cyanoacrylates_2021
Record Dates: First submitted 2022-06-27; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Tooth Socket
MeSH Terms: interventions — MK 6 cyanoacrylate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental)
  Interventions: Other: Cyanoacrylate glue
- Control group (Active Comparator)
  Interventions: Other: Platelet-rich fibrin (PRF)

INTERVENTIONS:
Other: Cyanoacrylate glue — 8 sockets that will be treated by immediate implant placement and sealed by a Cyanoacrylate glue.
  Arms: Study group
Other: Platelet-rich fibrin (PRF) — 8 sockets that will be treated by immediate implant placement and sealed by PRF.
  Arms: Control group

SUMMARY:
The health of peri-implant soft tissues is one of the most important aspects necessary for the long-term survival of dental implants. The importance of the peri-implant mucosal region lies in the need to establish a tight seal that isolates the implant and the bone from the oral environment. Study objective is to clinically compare the soft tissue healing, height, and thickness over immediate implants placed in type I sockets sealed by PRF to those sealed by a Cyanoacrylate glue.

DETAILED DESCRIPTION:
the study will be conducted on 16 extraction sockets in humans. Sockets will be randomly divided into two groups: Group I (test) will comprise 8 sockets sealed by PRF after immediate implant placement. Group II: (test) will comprise 8 sockets sealed by cyanoacrylate glue after immediate implant placement

ELIGIBILITY:
Inclusion Criteria:

* Any non-restorable hopeless tooth; a badly decayed tooth that cannot be restored, a Tooth with failed endodontic treatment, and tooth with longitudinal fracture.
* Post-extraction sockets type 1 with all bony walls intact; Type I extraction sockets according to Elian classification in 2007 have an intact labial plate of the bone and no soft tissue recession. Therefore, it does not require a mucoperiosteal flap elevation, only bone graft particles are packed into the socket after atraumatic extraction and socket debridement, then sealed with barrier membranes or soft tissue graft
* A good standard of oral hygiene.
* No signs of active periodontal disease in the selected tooth.

Exclusion Criteria:

* The presence of any systemic disease that could complicate bone or soft tissue healing after immediate implant placement.
* The presence of Acute periapical infection.
* The presence of any local factor that may interfere with extraction as tooth ankyloses. (
* Subjects who had undergone therapeutical radiation. (38)
* Patients who had been subjected to or who were under bisphosphonate therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in soft tissue healing | at 2nd week and 4th week
  Soft tissue healing will be assessed in both groups in reference to the soft tissue healing index according to Landry index Landry index scores
  Very poor: Tissue color: ≥50% of gingiva red Response to palpation: BleedingGranulation tissue: PresentIncision margin: Not epithelialized, with loss of epithelium beyond incision marginSuppuration: Present
  Poor: Tissue color: ≥50% of gingiva red Response to palpation: BleedingGranulation tissue: PresentIncision margin: Not epithelialized, with connective tissue exposed
  Good: Tissue colour: ≥25% and<50% of gingiva redResponse to palpation: No bleedingGranulation tissue: NoneIncision margin: No connective tissue exposed
  Very good: Tissue colour: <25% of gingiva redResponse to palpation: No bleedingGranulation tissue: NoneIncision margin: No connective tissue exposed
  Excellent: Tissue color: All tissues pinkResponse to palpation: No bleedingGranulation tissue: NoneIncision margin: No connective tissue exposed
Change in Mid crestal soft tissue thickness | at baseline and after 4 weeks
  Mid crestal soft tissue thickness over the immediate implant will be measured using a periodontal probe passing through soft tissue in the intersection midpoint of both buccolingual and mesiodistal dimensions of the socket till cover screw, after 4 weeks postoperatively
change in Mid-buccal soft tissue height | at baseline and after 4 weeks
  Mid-buccal soft tissue height: will be measured from gingival margin to implant platform, at surgery time and 4 weeks postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt